CLINICAL TRIAL: NCT05785130
Title: The Effects of White Noise for Adult Patients' Sleep Quality in Intensive Care Unit: a Randomized Controlled Trial
Brief Title: The Effects of White Noise for Adult Patients' Sleep Quality in Intensive Care Unit.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Collaborators: Kaohsiung Medical University (Other)
Responsible Party: Principal Investigator, Ya-Ching, Nien, Principal Investigator, Chang Gung Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 202300153B0
Record Dates: First submitted 2023-03-14; First posted 2023-03-27 (Actual); Results first posted 2025-03-17 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Sleep
Keywords: sleep quality; sleep disturbance; intensive care unit; critically ill patient
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Parasomnias

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- white noise group (Experimental): Background noise at bedtime.
  Interventions: Other: white noise
- conventional treatment group (No Intervention): Treatment as usual.

INTERVENTIONS:
Other: white noise — Using sound machine for 3 days at bedtime for 7 hours(11p.m.- 6a.m.) in a decibel of 40-50.
  Arms: white noise group

SUMMARY:
Poor sleep quality is one of the most common problems among adult patients in the intensive care unit (ICU). The causes of sleep disturbance are complicated. Poor sleep quality can lead to negative consequences for patients' physical and mental health. Non-pharmacological interventions, such as white noise, have been recommended to increase the threshold level of sound during nighttime and achieve masking effects to improve subjective sleep quality. This study is a randomized controlled trial that compared two parallel patient groups.The hypothesis of this study is that white noise can improve sleep quality in adult ICU patients compared with conventional treatment group.

DETAILED DESCRIPTION:
Poor sleep quality is one of the most common problems among adult patients in the intensive care unit (ICU). Statistics indicate that over 50% of ICU patients report sleep abnormalities, such as sleep fragmentation, arousals, frequent awakenings, and poor sleep quality. The causes of sleep disturbance are complicated, with evidence suggesting that environmental factors such as noise, from alarms and machines that are active around the clock in the ICU, play a significant role. Poor sleep quality can lead to negative consequences for patients' physical and mental health.

Sleep promotion interventions, including both pharmacological and non-pharmacological approaches, have been proposed. However, the side effects of pharmacological intervention may also lead to poor outcomes. Therefore, non-pharmacological interventions, such as background noise, have been recommended to increase the threshold level of sound during nighttime and achieve masking effects to improve subjective sleep quality.

This study was conducted in randomized controlled trial that compared two parallel patient groups. Patients were included by convenience sampling in a medical center in Taiwan. The Verran and Snyder-Halpern Sleep Scale (VSHSS) was used to assess subjective sleep quality. The main purpose of this study was to investigate the effect of white noise intervention in sleep quality in adult intensive care unit patients.

ELIGIBILITY:
Inclusion Criteria:

* Age must be greater than or equal to 20 years old.
* Admitted to the ICU and have been intubated for at least 24 hours.
* Aware of people, time, and place, and without hearing impairment.
* Be able to communicate in writing.
* The Glasgow Coma Scale score must be equal to or greater than 11, with a vocal response of 1 in the patient post-endotracheal tube placement.

Exclusion Criteria:

* History of insomnia, Alzheimer's disease, or depression.
* Routine use of sedative-hypnotic drugs (opioids, benzodiazepines, non-benzodiazepines, antihistamines, and melatonin) before admission.
* Post-operation in the operating room before ICU admission.
* ICDSC score of at least 4 or CAM-ICU positive.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-04-17 (Actual); Primary Completion 2024-08-04 (Actual); Study Completion 2024-11-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ya-Ching Nien, Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Chang Gung Memorial Hospital, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at in a medical center at southern Taiwan from March 2023 to August 2024.
Pre-assignment Details: Of 60 enrolled participants, 60 meets inclusion criteria and were randomized to white noise or conventional treatment group
Groups:
- White Noise Group: white noise at bedtime.
  white noise: Using sound machine for 3 days at bedtime for 7 hours(11p.m.- 6a.m.) in a decibel of 40-50.
- Conventional Treatment Group: Treatment as usual without white noise intervention
Period: Overall Study
Arm/Group | White Noise Group | Conventional Treatment Group
Started | 30 | 30
Completed | 29 (one of the participatants was withdrawl) | 29 (one of the participants on ECMO)
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Lack of Efficacy | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Conventional Treatment Group: Treatment as usual. without white nose intervention.
- Total: Total of all reporting groups
Arm/Group | White Noise Group | Conventional Treatment Group | Total
Number analyzed (Participants) | 29 | 29 | 58
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.76 (11.07) | 59.69 (15.74) | 61.72 (13.24)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 10 | 25
  Male | 14 | 19 | 33
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
APACHE II [Mean (Standard Deviation); unit: units on a scale] — The APACHE II (Acute Physiology and Chronic Health Evaluation II) score ranges from 0 to 71.
  The minimum score: 0 (indicating the least severe condition, with no acute physiological abnormalities or chronic health problems).
  The maximum score: 71 (indicating the most severe condition, with significant acute physiological abnormalities and severe chronic health problems).
  units on a scale | 20.41 (4.05) | 21.48 (5.77) | 20.95 (4.97)
comorbidity [Mean (Standard Deviation); unit: number of comorbidities] — The comorbility means one or more diseases that exist at the same times in one person.
  number of comorbidities | 1.66 (0.94) | 1.59 (1.30) | 1.62 (1.12)
Critical Care Pain Observation Tool(CPOT) [Mean (Standard Deviation); unit: scores on a scale] — The Critical Care Pain Observation Tool (CPOT) rates critically ill patients' pain based on clinical observation.
  The Critical Care Pain Observation Tool (CPOT) includes four observation indicators: facial expression, body movements, muscle tension, and ventilation (for ventilated patients). Each indicator is rated on a scale from 0 to 2 and the total score is obtained by adding the scores from each indicator. The total score of the CPOT range from 0 to 8 with a higher score indicating a higher level of pain.
  scores on a scale | 0.45 (0.87) | 0.83 (1.20) | 0.64 (1.05)
Education years [Mean (Standard Deviation); unit: years] | 10.62 (3.24) | 10.72 (3.28) | 10.67 (3.24)
Use painkiller [Count of Participants; unit: Participants]
  Yes | 9 | 12 | 21
  No | 20 | 17 | 37
Use hypnotic [Count of Participants; unit: Participants]
  Yes | 3 | 1 | 4
  No | 26 | 28 | 54

OUTCOME MEASURES:

1. Primary Outcome: The Verran and Snyder-Halpern Sleep Scale Scores on Baseline, the First Intervention Day(T1), the Third Intervention Day(T2), and Follow up Two Days Later After Intervention (T3) Between Two Groups.
Description: Sleep quality is assessed using the Verran and Snyder-Halpern (VSH) Sleep Scale, a subjective sleep scale that contains three dimensions: sleep disturbance, sleep effectiveness, and sleep supplementation, with a total of 15 items. Scores are measured using a visual analogue scale, which is a 100mm horizontal line. The maximum score is 100, and the minimum score is 0. The total score of the VSH Sleep Scale (VSHSS) ranges from 0 to 1500. The subscales are combined by summing the individual scores for each item, and the total score is obtained by adding the scores from each of the subscales. The lower the score, the poorer the sleep quality. Outcomes were measured at baseline, the first intervention day (T1), the third intervention day (T2), and two days after the intervention (T3) for both groups.
Time Frame: Baseline, 1st days, 3rd days and 5th days.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | White Noise Group | Conventional Treatment Group
Number analyzed (Participants) | 29 | 29
score on a scale
  baseline(T0) | 873.38 (262.24) | 898.45 (312.80)
  the first intervention day(T1) | 880.48 (226.89) | 746.91 (323.38)
  the third intervention day (T2) | 901.84 (259.23) | 665.91 (300.58)
  two days after the intervention (T3) | 774.17 (277.87) | 559.99 (268.25)
Statistical Analysis 1: Comparison: White Noise Group vs Conventional Treatment Group; It was calculated that 58 participants were randomized in a 1:1 between two arms on baseline, the first intervention day(T1), the third intervention day(T2), and follow up two days later after intervention (T3) . Sample size was determoned using G-power repeated measures, between factors(α = 0.05, power = 0.8). Assumption a discontinution rate of 10%; Test type: Superiority — T0; p = 0.74, t-test, 2 sided — T0; Mean Difference (Final Values) = -25.07
Statistical Analysis 2: Comparison: White Noise Group vs Conventional Treatment Group; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.75, t-test, 2 sided — T1; Median Difference (Final Values) = 133.57
Statistical Analysis 3: Comparison: White Noise Group vs Conventional Treatment Group; [analysis description as in outcome 1, analysis 1]; Test type: Superiority — T; p < 0.01, t-test, 2 sided — T2; Median Difference (Final Values) = 235.93
Statistical Analysis 4: Comparison: White Noise Group vs Conventional Treatment Group; [analysis description as in outcome 1, analysis 1]; Test type: Superiority — T3; p < 0.01, t-test, 2 sided — T3; Median Difference (Final Values) = 214.18

ADVERSE EVENTS:
Time Frame: 5 days
Groups:
- Conventional Treatment Group: Treatment as usual without whote noise intervention.
Arm/Group | White Noise Group | Conventional Treatment Group
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/29
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/29
Other Adverse Events (participants affected / at risk) | 0/29 | 0/29

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-03-02): https://cdn.clinicaltrials.gov/large-docs/30/NCT05785130/Prot_SAP_000.pdf